CLINICAL TRIAL: NCT03225742
Title: The Impact of Postoperative Catheterization Time After Stress Incontinence Surgery to Voiding Dysfunction, Urinary Retention and Success of Surgery
Brief Title: The Impact of Postoperative Catheterization Time After Stress Incontinence Surgery to Success of Surgery
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kerem Doga Seckin, ass prof, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2016/01
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2018-03

CONDITIONS: Stress Urinary Incontinence; Surgery
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- urinary catheterization time; one day: the patient urinary catheterization after surgery; one day
  Interventions: Diagnostic Test: to measure the residual volume after catheterization
- urinary catheterization time; two day: the patient urinary catheterization after surgery; two day
  Interventions: Diagnostic Test: to measure the residual volume after catheterization

INTERVENTIONS:
Diagnostic Test: to measure the residual volume after catheterization — after first micturition to measure the residual volume in bladder

SUMMARY:
After incontinence surgery, the patients randomly will be divided two groups. In group A postoperative urinary catheterization time will be applied one day, In group B catheterization will be applied two days. After removal of urinary catheter, residual volume will be measured and voiding function will be controlled. In postoperative period; third, sixth month and one year after surgery stress test will be applied to control success of surgery

ELIGIBILITY:
Inclusion Criteria:

* stress incontinence
* resistant to medical treatment

Exclusion Criteria:

* had no surgery before
* has no accompanying uterine descensus
* has no neurogenic disorder

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: the women who have stress incontinence at physical examination and urodynamics tests
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
early postoperative voiding dysfunction and urinary retention | two days
  after removal of urinary catheter, has residual volume much more than 150cc (to be measured with urinary catheterization)

SECONDARY OUTCOMES:
The success of stress urinary incontinence surgery | third month, sixth month and one year
  third, sixth month and one year after surgery, absence of stress urinary incontinence

CONTACTS AND LOCATIONS:
Locations (1):
- Kerem Doga Seckin, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No